CLINICAL TRIAL: NCT01880177
Title: A Study Designed to Develop and Validate a New Screening Measure for Identifying Undiagnosed At-Risk COPD Cases
Brief Title: Developing a COPD Case Finding Methodology for Primary Care
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: United BioSource, LLC (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Fernando J. Martinez, MD, MS, Professor, Department of Internal Medicine at University of Michigan, University of Michigan
Other Study IDs: HUM00068783; 7R01HL114055-03 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-18 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Current smokers: Current smokers (>10 pk yrs.)
- Ex-smokers: Ex-smokers with a history of >10 pk yrs
- Never-smokers: Never-smokers, defined as ≤100 cigarettes/pipes/cigars over life

SUMMARY:
The purpose of this qualitative work is to inform the content and structure of a new screening measure for identifying undiagnosed at-risk COPD cases in primary care and support content validity of the measure. This work will build on the results of a comprehensive literature review and data mining analyses by identifying the symptomatic and health event experiences of at-risk and newly diagnosed patients, as described by the patients themselves. Specific objectives are as follows:

Objective 1: To elicit concepts and symptom descriptions of COPD from patients with a recent diagnosis of COPD and those without a diagnosis but with risk factors for the disease. The qualitative information obtained in these focus groups will be used to develop a new questionnaire for identifying undiagnosed at-risk COPD cases in various clinic settings.

Objective 2: To review the new questionnaire with a new set of participants with a recent COPD diagnosis or those at risk for COPD to ensure that: (a) the instructions are clear, (b) the content of each question is appropriate and understandable to participants, (c) the intended connotation of each questions is consistent with participants' interpretation or assigned meaning, and (d) to assure that content is not seen as redundant across items. This will be done through one-on-one cognitive interviews.

Objective 3: To gather data on the ease/difficulty of peak flow meter use by people without or with a new diagnosis of COPD and the consistency of readings between electronic and mechanical readings in these patients. This information will be used to inform the development of peak-flow meter instructions for use as part of the screening methodology.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥40 years
* 2. Current smokers (>10 pk yrs.) or Ex-smokers with a history of >10 pk yrs. or Never-smokers, defined as ≤100 cigarettes/pipes/cigars over life
* 3. Stable state PFT values from within the last 12 months available or obtainable
* 4. Willing and able to attend the focus group session or cognitive interview
* 5. Able to read and speak in English
* 6. Willing and able to provide written Informed Consent

Exclusion Criteria:

* 1. Cognitive impairment, hearing or sight difficulty, or severe psychopathology that could interfere with ability to participate in the study
* 2. Patient was hospitalized for respiratory infection within the past 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through multiple clinic settings, i.e., pulmonology clinics, internal medicine clinics, and primary care/family medicine clinics.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
COPD Case Finding Tool | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, MS, Principal Investigator — University of Michigan; Nancy K Leidy, PhD, Principal Investigator — United BioSource, LLC; David Mannino, MD, Principal Investigator — University of Kentucky
Locations (4):
- United States (4):
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - UNMC College of Medicine, Omaha, Nebraska
  - Columbia University Medical center / New York Presbyterian Hospital, New York, New York

REFERENCES:
- [Background] Mannino DM, Homa DM, Akinbami LJ, Ford ES, Redd SC. Chronic obstructive pulmonary disease surveillance--United States, 1971-2000. Respir Care. 2002 Oct;47(10):1184-99. PMID 12354338
- [Background] Centers for Disease Control and Prevention (CDC). Deaths from chronic obstructive pulmonary disease--United States, 2000-2005. MMWR Morb Mortal Wkly Rep. 2008 Nov 14;57(45):1229-32. PMID 19008792
- [Background] Brown DW, Croft JB, Greenlund KJ, Giles WH. Trends in hospitalization with chronic obstructive pulmonary disease-United States, 1990-2005. COPD. 2010 Feb;7(1):59-62. doi: 10.3109/15412550903499548. PMID 20214464
- [Background] Mannino DM, Gagnon RC, Petty TL, Lydick E. Obstructive lung disease and low lung function in adults in the United States: data from the National Health and Nutrition Examination Survey, 1988-1994. Arch Intern Med. 2000 Jun 12;160(11):1683-9. doi: 10.1001/archinte.160.11.1683. PMID 10847262
- [Background] Anzueto A, Sethi S, Martinez FJ. Exacerbations of chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2007 Oct 1;4(7):554-64. doi: 10.1513/pats.200701-003FM. PMID 17878469
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Background] Roche N, Gaillat J, Garre M, Meunier JP, Lemaire N, Bendjenana H. Acute respiratory illness as a trigger for detecting chronic bronchitis in adults at risk of COPD: a primary care survey. Prim Care Respir J. 2010 Dec;19(4):371-7. doi: 10.4104/pcrj.2010.00042. PMID 20842324
- [Background] Langsetmo L, Platt RW, Ernst P, Bourbeau J. Underreporting exacerbation of chronic obstructive pulmonary disease in a longitudinal cohort. Am J Respir Crit Care Med. 2008 Feb 15;177(4):396-401. doi: 10.1164/rccm.200708-1290OC. Epub 2007 Nov 29. PMID 18048806
- [Background] Gruffydd-Jones K, Loveridge C. The 2010 NICE COPD Guidelines: how do they compare with the GOLD guidelines? Prim Care Respir J. 2011 Jun;20(2):199-204. doi: 10.4104/pcrj.2011.00011. PMID 21437566
- [Background] Wilt TJ, Niewoehner D, MacDonald R, Kane RL. Management of stable chronic obstructive pulmonary disease: a systematic review for a clinical practice guideline. Ann Intern Med. 2007 Nov 6;147(9):639-53. doi: 10.7326/0003-4819-147-9-200711060-00009. PMID 17975187
- [Background] Postma D, Anzueto A, Calverley P, Jenkins C, Make BJ, Sciurba FC, Similowski T, van der Molen T, Eriksson G. A new perspective on optimal care for patients with COPD. Prim Care Respir J. 2011 Jun;20(2):205-9. doi: 10.4104/pcrj.2011.00041. PMID 21559550
- [Background] Albert RK, Connett J, Bailey WC, Casaburi R, Cooper JAD, Criner GJ, Curtis JL, Dransfield MT, Han M, Lazarus SC, Make B, Marchetti N, Martinez FJ, Madinger NE, McEvoy C, Niewoehner DE, Porsasz J, Price CS, Reilly J, Scanlon PD, Sciurba FC, Scharf SM, Washko GR, Woodruff PG, and Anthonisen NR for the COPD Clinical Research Network. Chronic Administration of Azithromycin Decreases the Frequency of Chronic Obstructive Pulmonary Disease Exacerbations. Results of a Randomized Trail. NEJM 2011. In Press.
- [Background] Wilt TJ, Niewoehner D, Kim C, Kane RL, Linabery A, Tacklind J, Macdonald R, Rutks I. Use of spirometry for case finding, diagnosis, and management of chronic obstructive pulmonary disease (COPD). Evid Rep Technol Assess (Summ). 2005 Aug;(121):1-7. doi: 10.1037/e439492005-001. No abstract available. PMID 16238364
- [Background] Van Schayck CP, Loozen JM, Wagena E, Akkermans RP, Wesseling GJ. Detecting patients at a high risk of developing chronic obstructive pulmonary disease in general practice: cross sectional case finding study. BMJ. 2002 Jun 8;324(7350):1370. doi: 10.1136/bmj.324.7350.1370. PMID 12052807
- [Background] Freeman D, Nordyke RJ, Isonaka S, Nonikov DV, Maroni JM, Price D, Halbert RJ. Questions for COPD diagnostic screening in a primary care setting. Respir Med. 2005 Oct;99(10):1311-8. doi: 10.1016/j.rmed.2005.02.037. Epub 2005 Apr 18. PMID 16140231
- [Background] Price DB, Tinkelman DG, Halbert RJ, Nordyke RJ, Isonaka S, Nonikov D, Juniper EF, Freeman D, Hausen T, Levy ML, Ostrem A, van der Molen T, van Schayck CP. Symptom-based questionnaire for identifying COPD in smokers. Respiration. 2006;73(3):285-95. doi: 10.1159/000090142. Epub 2005 Dec 5. PMID 16330875
- [Background] Tinkelman DG, Price DB, Nordyke RJ, Halbert RJ, Isonaka S, Nonikov D, Juniper EF, Freeman D, Hausen T, Levy ML, Ostrem A, van der Molen T, van Schayck CP. Symptom-based questionnaire for differentiating COPD and asthma. Respiration. 2006;73(3):296-305. doi: 10.1159/000090141. Epub 2005 Dec 5. PMID 16330874
- [Background] Price DB, Tinkelman DG, Nordyke RJ, Isonaka S, Halbert RJ; COPD Questionnaire Study Group. Scoring system and clinical application of COPD diagnostic questionnaires. Chest. 2006 Jun;129(6):1531-9. doi: 10.1378/chest.129.6.1531. PMID 16778271
- [Background] Kotz D, Nelemans P, van Schayck CP, Wesseling GJ. External validation of a COPD diagnostic questionnaire. Eur Respir J. 2008 Feb;31(2):298-303. doi: 10.1183/09031936.00074307. Epub 2007 Oct 24. PMID 17959636
- [Background] Martinez FJ, Raczek AE, Seifer FD, Conoscenti CS, Curtice TG, D'Eletto T, Cote C, Hawkins C, Phillips AL; COPD-PS Clinician Working Group. Development and initial validation of a self-scored COPD Population Screener Questionnaire (COPD-PS). COPD. 2008 Apr;5(2):85-95. doi: 10.1080/15412550801940721. PMID 18415807
- [Background] Yawn BP, Mapel DW, Mannino DM, Martinez FJ, Donohue JF, Hanania NA, Kosinski M, Rendas-Baum R, Mintz M, Samuels S, Dalal AA; Lung Function Questionnaire Working Group. Development of the Lung Function Questionnaire (LFQ) to identify airflow obstruction. Int J Chron Obstruct Pulmon Dis. 2010 Feb 18;5:1-10. PMID 20368906
- [Background] Hanania NA, Mannino DM, Yawn BP, Mapel DW, Martinez FJ, Donohue JF, Kosinski M, Rendas-Baum R, Mintz M, Samuels S, Jhingran P, Dalal AA. Predicting risk of airflow obstruction in primary care: Validation of the lung function questionnaire (LFQ). Respir Med. 2010 Aug;104(8):1160-70. doi: 10.1016/j.rmed.2010.02.009. Epub 2010 Mar 11. PMID 20226647
- [Background] Frith P, Crockett A, Beilby J, Marshall D, Attewell R, Ratnanesan A, Gavagna G. Simplified COPD screening: validation of the PiKo-6(R) in primary care. Prim Care Respir J. 2011 Jun;20(2):190-8, 2 p following 198. doi: 10.4104/pcrj.2011.00040. PMID 21597667
- [Background] Sichletidis L, Spyratos D, Papaioannou M, Chloros D, Tsiotsios A, Tsagaraki V, Haidich AB. A combination of the IPAG questionnaire and PiKo-6(R) flow meter is a valuable screening tool for COPD in the primary care setting. Prim Care Respir J. 2011 Jun;20(2):184-9, 1 p following 189. doi: 10.4104/pcrj.2011.00038. PMID 21597666
- [Background] Patrick DL, Burke LB, Powers JH, Scott JA, Rock EP, Dawisha S, O'Neill R, Kennedy DL. Patient-reported outcomes to support medical product labeling claims: FDA perspective. Value Health. 2007 Nov-Dec;10 Suppl 2:S125-37. doi: 10.1111/j.1524-4733.2007.00275.x. PMID 17995471
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Leidy NK, Vernon M. Perspectives on patient-reported outcomes : content validity and qualitative research in a changing clinical trial environment. Pharmacoeconomics. 2008;26(5):363-70. doi: 10.2165/00019053-200826050-00002. PMID 18429654
- [Derived] Leidy NK, Martinez FJ, Malley KG, Mannino DM, Han MK, Bacci ED, Brown RW, Houfek JF, Labaki WW, Make BJ, Meldrum CA, Quezada W, Rennard S, Thomashow B, Yawn BP. Can CAPTURE be used to identify undiagnosed patients with mild-to-moderate COPD likely to benefit from treatment? Int J Chron Obstruct Pulmon Dis. 2018 Jun 13;13:1901-1912. doi: 10.2147/COPD.S152226. eCollection 2018. PMID 29942123
- [Derived] Quezada WA, Whippo BA, Jellen PA, Leidy NK, Mannino DM, Kim KJ, Han MK, Houfek JF, Make B, Malley KG, Meldrum CA, Rennard SI, Yawn BP, Martinez FJ, Thomashow BM; High-Risk-COPD Screening Study Group( *). How Well Does CAPTURE Translate?: An Exploratory Analysis of a COPD Case-Finding Method for Spanish-Speaking Patients. Chest. 2017 Oct;152(4):761-770. doi: 10.1016/j.chest.2017.03.047. Epub 2017 Apr 14. PMID 28414029
- [Derived] Martinez FJ, Mannino D, Leidy NK, Malley KG, Bacci ED, Barr RG, Bowler RP, Han MK, Houfek JF, Make B, Meldrum CA, Rennard S, Thomashow B, Walsh J, Yawn BP; High-Risk-COPD Screening Study Group *. A New Approach for Identifying Patients with Undiagnosed Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Mar 15;195(6):748-756. doi: 10.1164/rccm.201603-0622OC. PMID 27783539